CLINICAL TRIAL: NCT00475969
Title: Duloxetine Hydrochloride Once Daily Compared With Placebo in the Treatment of Generalized Anxiety Disorder
Brief Title: Duloxetine vs Placebo in the Treatment of General Anxiety
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6089; F1J-MC-HMDT
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Last update posted 2007-05-21 (Estimated); Status verified 2007-05

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: duloxetine
Drug: placebo

SUMMARY:
To see if duloxetine 60 to 120 mg once daily (QD) is better than placebo in the treatment of generalized anxiety disorder (GAD).

DETAILED DESCRIPTION:
duloxetine 60 to 120 mg once daily (QD) and placebo 11 weeks

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients at least 18 years of age presenting with generalized anxiety disorder (GAD) based on the disease diagnostic criteria The patient must suffer from GAD and not from an adjustment disorder or anxiety disorder not otherwise specified (NOS). Symptoms of GAD should not be situational in nature.
* Females of childbearing potential (not surgically sterilized and between menarche and 1 year postmenopause) who are not breastfeeding; test negative for pregnancy at the time of enrollment based on a urine pregnancy test; and agree to use a reliable method of birth control during the study and for 1 week following the last dose of study drug.
* Must have a Clinical Global Impressions of Severity (CGI-Severity) score of greater than or equal to 4 at Visit 1 and Visit 2.
* At Visit 1, patient must have a Covi Anxiety Scale (CAS) score of greater than or equal to 9, no item in the Raskin Depression Scale (RDS) may be greater than 3, and the CAS must be greater than the RDS.
* Must have a Hospital Anxiety and Depression Scale (HADS) anxiety subscale score of greater than or equal to 10 at Visit 1.

Exclusion Criteria:

* Any current and primary DSM-IV Axis I diagnosis other than GAD.

  * Patients diagnosed with or who have a history of major depressive disorder (MDD) within the past 6 months or
  * Patients diagnosed with or who have a history of Panic Disorder, Post-Traumatic Stress Disorder (PTSD), or an eating disorder within the past year or
  * Patients who have been diagnosed with Obsessive Compulsive Disorder (OCD), Bipolar Affective Disorder, psychosis, factitious disorder, or somatoform disorders during their lifetime.
* The presence of an Axis II disorder or history of antisocial behavior, which, in the judgment of the investigator, would interfere with compliance with the study protocol.
* Benzodiazepine use 14 days prior to Visit 2.
* Patients judged clinically to be at serious suicidal risk, or patients who, in the opinion of the investigator, are poor medical or psychiatric risks for study completion.
* Have received treatment within the last 30 days with a drug (not including study drug) that has not received regulatory approval for any indication at the time of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327
Dates: Start 2004-08; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAMA) total score (Hamilton 1959)

SECONDARY OUTCOMES:
Sheehan Disability Scale (SDS) Global Functional Impairment score (Sheehan 1983)
Hospital Anxiety Depression Scale (HADS; Zigmond and Snaith 1983)
Clinical Global Impressions of Improvement scale (CGI-Improvement; Guy 1976)
Patient's Global Impressions of Improvement scale (PGI-Improvement; Guy 1976)
Symptom Questionnaire-Somatic Subscale (SQ-SS)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Sheehan DV, Harnett-Sheehan K, Spann ME, Thompson HF, Prakash A. Assessing remission in major depressive disorder and generalized anxiety disorder clinical trials with the discan metric of the Sheehan disability scale. Int Clin Psychopharmacol. 2011 Mar;26(2):75-83. doi: 10.1097/YIC.0b013e328341bb5f. PMID 21102344
- [Derived] Hartford JT, Endicott J, Kornstein SG, Allgulander C, Wohlreich MM, Russell JM, Perahia DG, Erickson JS. Implications of pain in generalized anxiety disorder: efficacy of duloxetine. Prim Care Companion J Clin Psychiatry. 2008;10(3):197-204. doi: 10.4088/pcc.v10n0304. PMID 18615176
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com